CLINICAL TRIAL: NCT01421498
Title: A Phase 3, Multicenter, Randomized, Double- Masked and Placebo-Controlled Study Evaluating the Efficacy of a 5.0% Concentration of SAR 1118 Ophthalmic Solution Compared to Placebo in Subjects With Dry Eye (OPUS-1)
Brief Title: Safety and Efficacy Study of SAR 1118 to Treat Dry Eye Conducted in a Controlled Adverse Environment (CAE) (OPUS-1)
Acronym: OPUS-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1118-KCS-200
Record Dates: First submitted 2011-08-17; First posted 2011-08-22 (Estimated); Results first posted 2017-02-24 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Keratoconjunctivitis Sicca; Dry Eye Disease
Keywords: ophthalmic delivery; Dry Eye
MeSH Terms: conditions — Keratoconjunctivitis Sicca; Dry Eye Syndromes | interventions — lifitegrast

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5.0% Lifitegrast (Experimental): Lifitegrast
  Interventions: Drug: Lifitegrast
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lifitegrast — Dosage Form: Ophthalmic Solution Dosage: 5.0% Frequency: BID Duration: 12 weeks
  Other Names: SAR 1118
  Arms: 5.0% Lifitegrast
Drug: Placebo — Dosage Form: Ophthalmic Solution Frequency: BID Duration: 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy of SAR 1118 Ophthalmic Solution (5.0%) compared to placebo in the treatment of Dry Eye. The safety and tolerability of SAR 1118 Ophthalmic Solution (5.0%) compared to placebo in subjects with dry eye when administered BID for 12 weeks will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to read, sign, and date the informed consent and HIPAA documents
* Willing and able to comply with all study procedures
* Be at least 18 years of age
* Patient-reported history of dry eye in both eyes
* Demonstrate a positive response when exposed to the Controlled Adverse Environment model
* A negative urine pregnancy test if female of childbearing potential and must use adequate birth control throughout the study period

Exclusion Criteria:

* Any ocular condition that, in the opinion of the Investigator, could affect study parameters including, but not limited to, active ocular infection, ocular inflammation, glaucoma, and/or diabetic retinopathy
* Unwilling to avoid wearing contact lenses for 7 days prior to and for duration of the study period
* Any blood donation or significant loss of blood within 56 days of Visit 1
* Any history of immunodeficiency disorder, positive HIV, hepatitis B, C, or evidence of acute active hepatitis A (anti-HAV IgM), or organ or bone marrow transplant.
* Use of any topical ophthalmic preparations (including artificial tear substitutes) 72 hrs prior to Visit 1 and during the study
* Any significant chronic illness that could interfere with study parameters
* History of laser-assisted in situ keratomileusis (LASIK) or similar type of corneal refractive surgery within 12 months prior to Visit 1, and/or any other ocular surgical procedure within 12 months prior to Visit 1; or any scheduled ocular surgical procedure during the study period.
* Known history of alcohol and/or drug abuse
* Subjects with Dry eye secondary to scarring or destruction of conjunctival goblet cells (as with Vitamin A deficiency)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 588 (Actual)
Dates: Start 2011-08-29 (Actual); Primary Completion 2012-04-28 (Actual); Study Completion 2012-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (13):
- United States (13):
  - OPUS-1 Investigational Site, Waterbury, Connecticut
  - OPUS-1 Investigational Site, Louisville, Kentucky
  - OPUS-1 Investigational Site, Augusta, Maine
  - OPUS-1 Investigational Site, Lewiston, Maine
  - OPUS-1 Investigational Site, Andover, Massachusetts
  - OPUS-1 Investigational Site, Lancaster, Massachusetts
  - OPUS-1 Investigational Site, Quincy, Massachusetts
  - OPUS-1 Investigational Site, Wakefield, Massachusetts
  - OPUS-1 Investigational Site, Winchester, Massachusetts
  - OPUS-1 Investigational Site, Derry, New Hampshire
  - OPUS-1 Investigational Site, Manchester, New Hampshire
  - OPUS-1 Investigational Site, Memphis, Tennessee
  - OPUS-1 Investigational Site, Norfolk, Virginia

REFERENCES:
- [Result] Sheppard JD, Torkildsen GL, Lonsdale JD, D'Ambrosio FA Jr, McLaurin EB, Eiferman RA, Kennedy KS, Semba CP; OPUS-1 Study Group. Lifitegrast ophthalmic solution 5.0% for treatment of dry eye disease: results of the OPUS-1 phase 3 study. Ophthalmology. 2014 Feb;121(2):475-83. doi: 10.1016/j.ophtha.2013.09.015. Epub 2013 Nov 26. PMID 24289915

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted in a Controlled Adverse Environment (CAE).
Period: Overall Study
Arm/Group | Lifitegrast 5.0% | Placebo
Started | 293 | 295
Completed | 281 | 284
Not Completed | 12 | 11

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least 1 dose of investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifitegrast 5.0% | Placebo | Total
Number analyzed (Participants) | 293 | 295 | 588
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (12.21) | 61.1 (11.77) | 60.6 (11.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 229 | 217 | 446
  Male | 64 | 78 | 142

OUTCOME MEASURES:

1. Primary Outcome: Ocular Sign: Change From Baseline in Inferior Corneal Fluorescein Staining to Day 84
Description: Corneal staining was performed to grade the degree of corneal epithelial cell injury as measured by fluorescence using slit-lamp examination. The staining was graded with the Ophthalmic Research Associates, Inc. (ORA) scale. The corneal surface is divided into three regions: superior, central and inferior. The scores for each of these 3 regions ranged from 0 to 4 (0=no staining/none; 1=occasional/trace; 2=countable/mild; 3=uncountable, but not confluent/moderate; 4=confluent/severe) with 0.5 point increments, and lower score indicates a better outcome. Inferior corneal fluorescein staining scores from the study eye only were reported. Study eye is the 'worse eye', defined as the eye with worse (higher) score at baseline.
Time Frame: Baseline (Day 0) to Day 84
Population: Intent-to-Treat (ITT) population with Last Observation Carried Forward (LOCF) included all randomized participants who received at least 1 dose of investigational product.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifitegrast 5.0% | Placebo
Number analyzed (Participants) | 293 | 295
units on a scale | -0.07 (0.868) | 0.17 (0.819)
Statistical Analysis 1: Comparison: Lifitegrast 5.0% vs Placebo; Test type: Superiority or Other; p = 0.0007, t-test, 2 sided; Treatment difference = 0.24, 95% CI 2-sided [0.10 to 0.38]

2. Primary Outcome: Ocular Symptom: Change From Baseline in Visual-Related Subscale of the Symptom Functional Scale Score to Day 84
Description: The symptom functional scale is a validated instrument for ocular surface diseases, measuring the ocular symptoms, vision-related function, and environmental triggers. The 12 items of the symptom functional scale questionnaire were graded on a scale of 0 (none of the time) to 4 (all of the time). The index consisted of 3 sub scales: symptoms (sensitivity to light, gritty sensation, pain, blurred vision, and poor vision [Items 1-5]), visual-related sub scale of the symptom functional scale (ability to read, drive at night, use a computer, watch television [Items 6-9]), and environmental triggers (windy conditions, low humidity, air conditioning [Items 10-12]). The symptom functional scale was scored on a scale of 0 to 100, with higher scores representing greater disability. Negative change from baseline indicates improvement.
Time Frame: Baseline (Day 0) to Day 84
Population: ITT population with LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifitegrast 5.0% | Placebo
Number analyzed (Participants) | 293 | 295
units on a scale | -0.11 (0.829) | -0.12 (0.762)
Statistical Analysis 1: Comparison: Lifitegrast 5.0% vs Placebo; Test type: Superiority or Other; p = 0.7860, t-test, 2 sided; Treatment difference = -0.02, 95% CI 2-sided [-0.15 to 0.11]

ADVERSE EVENTS:
Arm/Group | Lifitegrast 5.0% | Placebo
Serious Adverse Events (participants affected / at risk) | 5/293 | 2/295
Other Adverse Events (participants affected / at risk) | 160/293 | 40/295
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lifitegrast 5.0% (N=293) | Placebo (N=295)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Non-Cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Infectious peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lifitegrast 5.0% (N=293) | Placebo (N=295)
Visual acuity reduced (Eye disorders) | 14 (17) | 15 (18)
Instillation site irritation (General disorders) | 69 (70) | 12 (12)
Instillation site pain (General disorders) | 63 (63) | 11 (11)
Instillation site pruritus (General disorders) | 19 (19) | 6 (6)
Instillation site reaction (General disorders) | 50 (52) | 2 (2)
Dysgeusia (Nervous system disorders) | 39 (40) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicentre publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicentre Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.